CLINICAL TRIAL: NCT04624464
Title: Assessing the Impact of Antimicrobial Exposure and Infection Control Measures on the Spread of Vancomycin-resistant Enterococcus Faecium (VREf) - A Prospective Study
Brief Title: Assessing the Impact of Antimicrobial Exposure and Infection Control Measures on the Spread of VRE
Acronym: AEGON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Collaborators: University of Freiburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Lübeck (Other)
Responsible Party: Principal Investigator, Dr. med. Jörg Janne Vehreschild, Prof. Dr., University Hospital of Cologne
Other Study IDs: 19-1325
Record Dates: First submitted 2020-07-30; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: VRE Infection; Antibiotic Resistant Infection
Keywords: VRE; Infection Control Measures; Antimicrobial Stewardship

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Biospecimen Retention: Samples With DNA — Cohort 1 (VRE negative at inclusion) and 2 (VRE positive at inclusion): Collection of rectal swabs for further microbiological analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: VRE negative at admission: 150 patients meeting the following inclusion criteria:
  * ≥ 18 years
  * Patients with malignant primary disease and current inpatient admission to a normal ward with expected inpatient stay of at least 15 days
  * High risk of exposure to antibiotics during the stay
  * Written informed consent of the patient after clarification has been given
  Exclusion criteria:
  * Already known current or documented past colonisation or infection by VRE
  * Simultaneous participation in other studies is only an exclusion criterion if the other study explicitly excludes participation in observational studies or if the other study complicates the interpretation of the endpoints of AEGON (e.g. double-blind study on antibiotic use).
  Interventions: Other: Rectal swabs - microbiological analysis
- Cohort 2: VRE positive at admission: A total 20 known VREf-positive patients meeting the following inclusion criteria:
  * Intestinal VREf colonization already known at the time of admission (e.g. based on examinations during previous stays or in external facilities)
  * Accommodation in a single room or alternatively multi-bed room with single occupancy on standard wards
  * Expected stay of at least 7 days
  Interventions: Other: Rectal swabs - microbiological analysis; Other: Examination of patient room

INTERVENTIONS:
Other: Rectal swabs - microbiological analysis — Microbial analyses will be performed from the rectal swabs obtained.
Other: Examination of patient room — Only performed for cohort 2
  Groups: Cohort 2: VRE positive at admission

SUMMARY:
The AEGON study is a German multicenter, prospective observational study. The study consists of two parts, which are carried out at all participating study sites and include two different patient cohorts. Part 1 focuses on the collection and analysis of rectal swabs from newly admitted VREf-negative patients at high risk of nosocomial VREf acquisition. Moreover, patients included into this part of the study will undergo in-depth documentation of clinical data if an antibiotic therapy is administered. Initiated antibiotic therapies will then be assessed by an AMS board (Antimicrobial Stewardship Board). In Part 2, environmental investigations will be performed in newly occupied single rooms of previously known VREf-positive patients. In addition, rectal swabs will be collected and data on antibiotic exposure of these patients will be documented in order to correlate the VRE contamination burden of surfaces with the intestinal VREf-load and antibiotic exposure.

DETAILED DESCRIPTION:
Current studies show that Vancomycin-resistant Enterococci (VRE) have become increasingly widespread throughout Germany in recent years, especially E. faecium (VREf). Healthy individuals can come into contact with VREf in various ways, for example via the food chain, contaminated drinking water or animal contacts. A possibly caused low-grade colonisation of the gastrointestinal tract with VREf (so-called low-level colonisation) can remain undetected during hospital admission using routine screening methods. The AEGON study, based on the use of state-of-the-art molecular diagnostics and comprehensive clinical data collection, will provide a detailed analysis of the factors involved in the rapid spread of VREf. In addition, diagnostic detection limits of common screening methods are determined by the use of additional diagnostics such as enrichment culture or molecular VREf detection.

The study is a German multicenter, prospective observational study and consists of two parts, which are carried out at all participating study sites and include two different patient cohorts. Part 1 focuses on the collection and analysis of rectal swabs from newly admitted VRE-negative patients at high risk of nosocomial VREf acquisition. Moreover, patients included into this part of the study will undergo in-depth documentation of clinical data if an antibiotic therapy is administered. Initiated antibiotic therapies will then be assessed by an AMS board. In Part 2, environmental investigations will be performed in newly occupied single rooms of previously known VREf-positive patients. In addition, rectal swabs will be collected and data on antibiotic exposure of these patients will be documented in order to correlate the VRE contamination burden of surfaces with the intestinal VREf-load and antibiotic exposure. The AEGON study, based on the use of state-of-the-art molecular diagnostics and comprehensive clinical data collection, will provide a detailed analysis of the factors involved in the rapid spread of VREf. In addition, diagnostic detection limits of common screening methods are determined by the use of additional diagnostics such as enrichment culture or molecular VREf detection.

ELIGIBILITY:
Part 1

Inclusion Criteria:

* ≥ 18 years
* Patients with malignant primary disease and current inpatient admission to a normal ward with expected inpatient stay of at least 15 days
* High risk of exposure to antibiotics during the stay
* Written informed consent of the patient after clarification has been given

Exclusion Criteria:

* Already known current or documented past colonisation or infection by VRE
* Simultaneous participation in other studies is only an exclusion criterion if the other study explicitly excludes participation in observational studies or if the other study complicates the interpretation of the endpoints of AEGON (e.g. double-blind study on antibiotic use).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selection of patients to be included in Part 1 of the AEGON study is based on the risk stratification for the nosocomial acquisition of VREf performed in the CONTROL study.
  It is planned to include a total of 150 patients from the participating study centers in Part 1. Based on the results of the CONTROL study, it can be assumed that within the selected target group in approx. 11% there is already an VREf colonisation by direct culture at admission and in 15% of the cases (22 of 150 patients) a nosocomial acquisition of VREf by direct culture (see method part) can be determined. Patients with VREcolonization detected at admission are excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
VREf - Intestinal microbiota | Baseline
  Primary Outcome for Cohort 1: Rate of VREf intestinal colonization detected by enrichment culture or specific PCR at time of uptake not detected by standard culture methods
VREf - Patient rooms | Change from baseline spread to spread at 10 weeks.
  Primary Outcome for Cohort 2: Description of the spread of VREf in single rooms newly enrolled in known VREf-positive patients

SECONDARY OUTCOMES:
Standard culture VREf detection | baseline and every week up to 10 weeks max.
  Cohort 1: Quantitative detection limit of standard culture methods for VREf detection compared to enrichment culture and qPCR (quantitative polymerase chain reaction)
Antibiotics | baseline and every week up to 10 weeks max.
  Cohort 1: Identification of antibiotic classes that increase the risk of clonal expansion and subsequent domination by VREf. Domination by VREf is defined as the combination of cultural VREf detection from a sample and 16S rRNA (16S ribosomal ribonucleic acid) sequencing of the relative frequency of the Enterococcus genus over 30% as the most abundant genus in the sample.
Inadequately administered antibiotics | baseline and every week up to 10 weeks max.
  Cohort 1: Proportion of inadequately administered antibiotics, defined as unnecessary, too long, too broad or too high doses in patients who develop VREf domination (see definition above) compared to patients without VREf acquisition and patients with VREf acquisition but without domination.
Adequate antibiotic | baseline and every week up to 10 weeks max.
  Cohort 1: Rate of patients with no or adequate antibiotic therapy compared to patients with inadequate antibiotic therapy who develop a new colonization with VREf during the stay
Influence of antibiotic exposure duration | baseline and every week up to 10 weeks max.
  Cohort 1: Influence of antibiotic exposure duration on microbiota
Influence of antibiotic class | baseline and every week up to 10 weeks max.
  Cohort 1: Influence of antibiotic class on microbiota
VREf contamination | baseline at least every 72 hours up to max of 20 days.
  Cohort 2: Identification of high risk objects and surfaces for VREf contamination in patient rooms with known VREf-positive patients
Correlation of the antibiotic exposure | baseline at least every 72 hours up to max of 20 days.
  Cohort 2: Correlation of the antibiotic exposure of already known VREf-positive patients with the contamination load of objects and surfaces in the corresponding patient room.
Contamination load of objects | baseline at least every 72 hours up to max of 20 days.
  Cohort 2: Correlation of the relative proportion of enterococci in intestinal microbiota with the contamination load of objects and surfaces in the associated patient room
Cleaning quality | baseline at least every 72 hours up to max of 20 days.
  Cohort 2: Correlation of cleaning quality with the contamination load of VREf on objects and surfaces in rooms of known VRE-positive patients

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Janne Vehreschild, Prof. Dr. med, Principal Investigator — University Hospital of Cologne; Maria J.G.T. Vehreschild, Prof. Dr. med, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gastmeier P, Schroder C, Behnke M, Meyer E, Geffers C. Dramatic increase in vancomycin-resistant enterococci in Germany. J Antimicrob Chemother. 2014 Jun;69(6):1660-4. doi: 10.1093/jac/dku035. Epub 2014 Mar 9. PMID 24615816
- [Background] Liss BJ, Vehreschild JJ, Cornely OA, Hallek M, Fatkenheuer G, Wisplinghoff H, Seifert H, Vehreschild MJ. Intestinal colonisation and blood stream infections due to vancomycin-resistant enterococci (VRE) and extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBLE) in patients with haematological and oncological malignancies. Infection. 2012 Dec;40(6):613-9. doi: 10.1007/s15010-012-0269-y. Epub 2012 Jun 5. PMID 22665143
- [Background] Vehreschild MJGT, Haverkamp M, Biehl LM, Lemmen S, Fatkenheuer G. Vancomycin-resistant enterococci (VRE): a reason to isolate? Infection. 2019 Feb;47(1):7-11. doi: 10.1007/s15010-018-1202-9. Epub 2018 Sep 3. PMID 30178076
- [Background] Biehl LM, Higgins P, Wille T, Peter K, Hamprecht A, Peter S, Dorfel D, Vogel W, Hafner H, Lemmen S, Panse J, Rohde H, Klupp EM, Schafhausen P, Imirzalioglu C, Falgenhauer L, Salmanton-Garcia J, Stecher M, Vehreschild JJ, Seifert H, Vehreschild MJGT. Impact of single-room contact precautions on hospital-acquisition and transmission of multidrug-resistant Escherichia coli: a prospective multicentre cohort study in haematological and oncological wards. Clin Microbiol Infect. 2019 Aug;25(8):1013-1020. doi: 10.1016/j.cmi.2018.12.029. Epub 2019 Jan 12. PMID 30641228